CLINICAL TRIAL: NCT03521271
Title: Investigation Of Factors Affecting Hand Functions in Nonambulatory Patients With Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gülcan Altınok, Master Student, Hacettepe University
Other Study IDs: GO 17/307
Record Dates: First submitted 2018-04-19; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Upper limb; Hand functions; Performance; Grip Strength
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study, determining the factors affecting the hand functions of children with Duchenne Muscular Dystrophy who have lost their independent ambulatory ability and determining the effects on the overall upper extremity performance and quality of life of the determined factors.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is the most common neuromuscular disease seen in childhood. DMD is an X linked recessive disorder. DMD is characterized by complete or partial (<3%) deficiency of the cell membrane protein dystrophin.

Dystrophin deficiency results in a permanent deterioration of muscle fibers. This leads to a progressive decrease in muscle strength and functional abilities. The precise mechanism of how the defect of dystrophin leads to degeneration of muscle fibers remains uncertain, but cytoskeletal deterioration, sarcolemmal instability and abnormal calcium homeostasis are thought to play a role in this degeneration.

These patients have symptoms such as limb proximals and progressive muscle weakness in the trunk, gait abnormalities, Gower's sign, various degrees of restriction in daily living activities, and frequent falls. The majority of patients have elevated serum creatine kinase or elevated liver transaminases and less frequently language or general developmental retardation.

Walking ability of this children begins to deteriorate between the ages of 3-6. These patients are generally dependent on wheelchair aged 10-12 years. The loss of walking is the milestone in terms of the progression of the disease. The use of electric wheelchairs limits arm functions such as lengthening and lifting during the late phase of the illness (when the ambulance has been lost and the ambulance is being continued with the wheelchair).

Patients with DMD have an average life span of 30 years with spinal surgery and ventilation support. They spend most of their lives dependent on the wheelchair and need functional use of the upper limbs to maintain the best possible level of independence in their daily life activities throughout their lifetimes.

Although muscle weakness in the proximal limbs is the first finding of the disease, the influence of upper extremity functions gives symptoms after 8 years of age and has a great influence on the level of independence of DMD patients in life since this process. For this reason, rehabilitation approaches for the protection of upper extremity functions from the early period of the disease are of great importance.Effective interventions are necessary to achieve this goal and these variables must be considered when making clinical decisions.

Patients with adult DMD have been shown to be able to perform important functional activities with limited distal motor function in the late phase of disease, but tend to lose these capacities as muscle strength decreases. For this reason, determining the factors (grip strength, thumb opposition, upper extremity joint range of motion, upper extremity muscle strength, etc.) that may affect hand functions, which is an important component in maintaining upper extremity functioning, and how these factors are related to the general functions of the upper extremity it is crucial that this disease leads to physiotherapy rehabilitation programs to be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Having a Duchenne Muscular Dystrophy diagnosis by a practicing physician,
* Between the ages of 8-16 years,
* Having lost ambulation ability,
* Brooke Upper Extremity Functional Classification (1-5)
* To have motivation and co-operation with physiotherapist for evaluations to be made

Exclusion Criteria:

* To maintain the capacity of independent ambulance,
* Having cooperative disorder or serious mental disorder,
* Any spinal and / or upper extremity injuries and / or surgery in the last 6 months,
* Having any systemic disease other than DMD,
* Not volunteering to participate in the study

Ages: 8 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who applied to the Pediatric Neuromuscular Diseases Unıt of Hacettepe University Physiotherapy and Rehabilitation Department
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Brooke Upper Extremity Functional Classification (1-6) | 2 minutes
  Children's functional levels were assessed with Brooke Upper Extremity Functional Classification (BUEFS) and children with a BUEFS score between 1-5 were included in the study.
  1. Starting with arms at sides, can abduct arms in a full circle until they touch above head
  2. Can raise arms above head only by flexing elbow or using accesory muscles
  3. Cannot raise arms above head but can raise a glass of water to mouth (using both hands if necessary)
  4. Can raise hands to mouth but cannot raise a glass of water to mouth
  5. Cannot raise hand to mouth but can use hands to hold pen or pick up pennies from table
  6. Cannot raise hands to mouth and has no useful function of hands
Passive joint range of motion | 10 minutes
  Passive range of motions were assessed with goniometer and recorded limitations.
Upper extremity muscle strength | 20 minutes
  Hand held dynamometer
Thumb opposition | 2 minutes
  Thumb opposition was assessed by Kapandji score (1-10). Score Location achieved
  1. Radial side of the proximal phalanx of the 2nd phalanx
  2. Radial side of the middle phalanx of the 2nd phalanx
  3. Tip of the 2nd phalanx
  4. Tip of the 3th phalanx
  5. Tip of the 4th phalanx
  6. Tip of the 5th phalanx
  7. Distal interphalangeal joint crease of the 5th phalanx
  8. Proximal interphalangeal joint crease of the 5th phalanx
  9. Metacarpophalangeal joint crease of the 5th phalanx
  10. Distal palmar crease
Lateral, tripod, two-point pinch strength | 3 minutes
  Pinchmeter
Performance of the upper extremity | 15 minutes
  Performance of the Upper Limb (PUL) (0-74) is including three dimension:
  * Shoulder dimension (0-16)
  * Elbow dimension (0-34)
  * Distal dimension (0-24)
Hand function | 3 minutes
  ABILHAND-Kids (0-36)
Activity limitations | 3 minutes
  ACTIVLIM (0-36)
Gross grip strength | 2 minutes
  Hand dynamometer

SECONDARY OUTCOMES:
Quality of life assessment of children (0-100) | 5 minutes
  PedsQL-Child report
Quality of life assessment of parents (0-100) | 5 minutes
  PedsQL-Parent report

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Samanpazarı/Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided